CLINICAL TRIAL: NCT02718898
Title: A Multicenter, Randomized, Double-Blind Study Comparing the Efficacy and Safety of Ixekizumab Versus Placebo in Patients With Moderate-to-Severe Genital Psoriasis
Brief Title: A Study of Ixekizumab (LY2439821) in Participants With Moderate-to-Severe Genital Psoriasis
Acronym: IXORA-Q
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16010; I1F-MC-RHBQ (Other: Eli Lilly and Company); 2015-002628-14 (EudraCT Number)
Record Dates: First submitted 2016-03-21; First posted 2016-03-24 (Estimated); Results first posted 2018-03-23 (Actual); Last update posted 2019-09-16 (Actual); Status verified 2019-08

CONDITIONS: Genital Psoriasis; Psoriasis
Keywords: genital
MeSH Terms: conditions — Psoriasis | interventions — ixekizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ixekizumab (Experimental): Blinded Treatment Period: 160 milligrams (mg) ixekizumab given subcutaneously (SC) at baseline followed by 80 mg ixekizumab every 2 weeks (Q2W) SC from week 2 to week 10. At week 12, 80 mg ixekizumab and placebo given SC.
  Open Label Period: 80 mg ixekizumab given SC every 4 weeks (Q4W) with an option for Q2W dosing starting at week 24, week 28 or week 40.
  Interventions: Drug: Ixekizumab; Drug: Placebo
- Placebo (Placebo Comparator): Blinded Treatment Period: Placebo given SC at baseline followed by placebo given SC Q2W from week 2 to week 10. At week 12, 160 mg ixekizumab given SC.
  Open Label Period: 80 mg ixekizumab given SC Q4W with an option for Q2W dosing starting at week 24, week 28 or week 40.
  Interventions: Drug: Ixekizumab; Drug: Placebo

INTERVENTIONS:
Drug: Ixekizumab — Administered SC
  Other Names: LY2439821
Drug: Placebo — Administered SC

SUMMARY:
The main purpose of this study is to evaluate the efficacy and safety of the study drug ixekizumab compared to placebo in participants with moderate-to-severe genital psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Have chronic plaque psoriasis based on a diagnosis of chronic plaque psoriasis for at least 6 months before baseline.
* Have moderate-to-severe psoriasis in the genital area at screening and baseline.
* Have plaque psoriasis in a nongenital area at screening and baseline.
* Have failed to respond to, or are intolerant of, at least 1 topical therapy used for treatment of psoriasis affecting the genital area.
* Must agree to use reliable method of birth control, which could include abstinence, during the study and for at least 12 weeks following the last dose of study drug.

Exclusion Criteria:

* Pustular, erythrodermic, and/or guttate forms of psoriasis.
* History of drug-induced psoriasis.
* Have recently received certain treatments for psoriasis (in particular, within the past 4 weeks but the restriction can go up to 12 months for some treatments).
* Have ever received treatment with ixekizumab, secukinumab, brodalumab, or another drug with a similar mode of action.
* Cannot avoid excessive sun exposure or use of tanning booths for at least 4 weeks prior to baseline and during the study.
* Are currently enrolled in any other clinical trial involving an investigational product.
* Serious disorder or illness other than plaque psoriasis.
* Active or history of malignant disease within 5 years prior to baseline.
* Serious infection within the last 3 months.
* Have received a live vaccine within 3 months of baseline or plan to do so during the study.
* Have received a vaccination with Bacillus Calmette-Guérin (BCG) within the past year.
* Pregnant or breastfeeding (lactating) women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2016-04; Primary Completion 2017-02-22 (Actual); Study Completion 2018-02-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (32):
- United States (13):
  - Southern California Dermatology, Santa Ana, California
  - Clinical Science Institute, Santa Monica, California
  - Olympian Clinical Research, Tampa, Florida
  - Advanced Medical Research, Sandy Springs, Georgia
  - Dawes Fretzin Clinical Research, Indianapolis, Indiana
  - The South Bend Clinic, South Bend, Indiana
  - Tufts Medical Center, Boston, Massachusetts
  - Oregon Medical Research Center, Portland, Oregon
  - Clinical Partners LLC, Johnston, Rhode Island
  - Modern Research Associates PLLC, Dallas, Texas
  - Menter Dermatology Research Institute, Dallas, Texas
  - Pflugerville Dermatology Clinical Research Center, Pflugerville, Texas
  - University of Utah, Salt Lake City, Utah
- Australia (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Adelaide
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Carlton
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Darlinghurst
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Woolloongabba
- Austria (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Graz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vienna
- Belgium (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brussels
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ghent
- Canada (5):
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., London
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Markham
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Montreal
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Québec
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Surrey
- Netherlands (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bergen op Zoom
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Breda
- GCM Medical Group PSC, San Juan, Puerto Rico
- Turkey (Türkiye) (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bursa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gaziantep
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Istanbul

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- See also: Click here for more information about this study: A Study of Ixekizumab (LY2439821) in Participants With Moderate-to-Severe Genital Psoriasis (IXORA-Q) — http://www.lillytrialguide.com/en-US/studies/genital-psoriasis/RHBQ#?postal=

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 12 week Blinded Treatment period, followed by 40 week Open Label Treatment Period, followed by 12 week Post treatment follow-up period.
  ttt = treatment, Pt = Participant.
Groups:
- Placebo - Blinded Treatment: Participants received placebo subcutaneously at baseline and every 2 weeks (Q2W) from week 2 to week 10. At week 12, 160 mg Ixekizumab was given by Subcutaneous injection during blinded treatment period.
- Ixekizumab 80mg Q2W - Blinded Treatment: Participants received 160 milligrams (mg) Ixekizumab subcutaneously (SC) at baseline followed by 80mg Ixekizumab every 2 weeks (Q2W) from week 2 to week 10. At week 12, 80mg Ixekizumab and placebo was given SC during blinded treatment period.
- Placebo/Ixekizumab 80mg Q4W - Open Label Treatment Period: Participants who received placebo in blinded treatment Period had received initial dose of 160mg Ixekizumab at week 12 followed by 80mg Ixekizumab Q4W by subcutaneous injection in open label treatment period.
  Participants had an option to step-up to Q2W dosing starting at week 24 through week 40.
- Ixekizumab 80mg Q2W/Ixekizumab 80mg Q4W - Open Label Treatment: Participants who received Ixekizumab in blinded treatment Period had received initial dose of 80mg Ixekizumab & placebo at week 12 followed by 80mg Ixekizumab Q4W by subcutaneous injection in open label treatment period.
  Participants had an option to step-up to Q2W dosing starting at week 24 through week 40.
- Placebo - Post Treatment Follow-up; Ixeqizumab 80mg Q4W - Post Treatment Follow-up Period; Ixekizumab 80mg Q2W - Post Treatment Follow-up: Participants did not receive any study treatment during post treatment follow-up period.
Period: Blinded Treatment Period
Arm/Group | Placebo - Blinded Treatment | Ixekizumab 80mg Q2W - Blinded Treatment | Placebo/Ixekizumab 80mg Q4W - Open Label Treatment Period | Ixekizumab 80mg Q2W/Ixekizumab 80mg Q4W - Open Label Treatment | Placebo - Post Treatment Follow-up | Ixeqizumab 80mg Q4W - Post Treatment Follow-up Period | Ixekizumab 80mg Q2W - Post Treatment Follow-up
Started | 74 | 75 | 0 | 0 | 0 | 0 | 0
Completed | 65 | 74 | 0 | 0 | 0 | 0 | 0
Not Completed | 9 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 5 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 2 | 0 | 0 | 0 | 0 | 0 | 0
Period: Open Label Treatment Period (OLTP)
Arm/Group | Placebo - Blinded Treatment | Ixekizumab 80mg Q2W - Blinded Treatment | Placebo/Ixekizumab 80mg Q4W - Open Label Treatment Period | Ixekizumab 80mg Q2W/Ixekizumab 80mg Q4W - Open Label Treatment | Placebo - Post Treatment Follow-up | Ixeqizumab 80mg Q4W - Post Treatment Follow-up Period | Ixekizumab 80mg Q2W - Post Treatment Follow-up
Started | 0 | 0 | 65 | 74 | 0 | 0 | 0
Completed | 0 | 0 | 62 | 64 | 0 | 0 | 0
Not Completed | 0 | 0 | 3 | 10 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 3 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 1 | 2 | 0 | 0 | 0
Not completed — Subject discontinued in OLTP | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Ttt of undisclosed addiction-Pt withdrew | 0 | 0 | 0 | 1 | 0 | 0 | 0
Period: Post Treatment Follow-up Period
Arm/Group | Placebo - Blinded Treatment | Ixekizumab 80mg Q2W - Blinded Treatment | Placebo/Ixekizumab 80mg Q4W - Open Label Treatment Period | Ixekizumab 80mg Q2W/Ixekizumab 80mg Q4W - Open Label Treatment | Placebo - Post Treatment Follow-up | Ixeqizumab 80mg Q4W - Post Treatment Follow-up Period | Ixekizumab 80mg Q2W - Post Treatment Follow-up
Started | 0 | 0 | 0 | 0 | 1 (One participant who discontinued from placebo blinded treatment had entered post-treatment follow-up) | 78 | 49
Completed | 0 | 0 | 0 | 0 | 0 | 67 | 44
Not Completed | 0 | 0 | 0 | 0 | 1 | 11 | 5
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 5 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 5 | 3

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Participants received placebo subcutaneously at baseline and every 2 weeks (Q2W) from week 2 to week 10. At week 12, 160 mg Ixekizumab given SC.
- Ixekizumab 80mg Q2W: Participants received 160 milligrams (mg) Ixekizumab subcutaneously (SC) at baseline followed by 80 mg Ixekizumab every 2 weeks (Q2W) from week 2 to week 10. At week 12, 80 mg Ixekizumab and placebo was given SC during blinded treatment period.
- Total: Total of all reporting groups
Arm/Group | Placebo | Ixekizumab 80mg Q2W | Total
Number analyzed (Participants) | 74 | 75 | 149
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.4 (12.55) | 43.1 (12.95) | 43.7 (12.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 19 | 36
  Male | 57 | 56 | 113
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 13 | 27
  Not Hispanic or Latino | 57 | 60 | 117
  Unknown or Not Reported | 3 | 2 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 7 | 3 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 64 | 67 | 131
  More than one race | 1 | 4 | 5
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 16 | 13 | 29
  Puerto Rico | 4 | 7 | 11
  Austria | 4 | 4 | 8
  Netherlands | 2 | 3 | 5
  Turkey | 3 | 4 | 7
  Belgium | 3 | 4 | 7
  United States | 31 | 31 | 62
  Australia | 11 | 9 | 20
sPGA of Genitalia [Mean (Standard Deviation); unit: units on a scale] — The Static Physician Global Assessment (sPGA) of Genitalia score is based on a combination of erythema and the secondary features (plaque elevation and/or scale). For the analysis of responses, the participant's psoriasis is assessed as follows: 0 = clear,1 = minimal,2 = mild,3 = moderate,4 = severe,5 = very severe.
  units on a scale | 3.5 (0.53) | 3.4 (0.61) | 3.4 (0.57)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Achieving Static Physician Global Assessment (sPGA) of Genitalia (0,1)
Description: sPGA of Genitalia score is based on a combination of erythema and the secondary features (plaque elevation and/or scale). For the analysis of responses, the participant's psoriasis was assessed as follows: 0 = clear,1 = minimal, 2 = mild, 3 = moderate, 4 = severe, 5 = very severe.
  sPGA of Genitalia (0,1) : A sPGA of Genitalia assessed as either 0 or 1.
Time Frame: Week 12
Population: All randomized participants.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: Participants received placebo subcutaneously at baseline and every 2 weeks (Q2W) from week 2 to week 10. At week 12, 160 mg Ixekizumab was given by subcutaneous injection.
Arm/Group | Placebo | Ixekizumab 80mg Q2W
Number analyzed (Participants) | 74 | 75
Participants | 6 | 55
Statistical Analysis 1: Comparison: Placebo vs Ixekizumab 80mg Q2W; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 33.80, 95% CI 2-sided [12.39 to 92.23]

2. Secondary Outcome: Number of Participants Achieving Overall sPGA (0,1)
Description: The overall sPGA is the physician's global assessment of the participant's psoriasis (Ps) lesions at a given time point. Plaques were assessed for induration, erythema, and scaling, and an overall rating of psoriasis severity was given using the anchors of 0 = clear, 1 = minimal, 2 = mild, 3 = moderate, 4 = severe, 5 = very severe.
  Overall sPGA (0,1) : An overall sPGA assessed as either 0 or 1.
Time Frame: Week 12
Population: All randomized participants.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: Participants received placebo subcutaneously at baseline and every 2 weeks (Q2W) from week 2 to week 10. At week 12, 160 mg Ixekizumab was by given subcutaneous injection.
Arm/Group | Placebo | Ixekizumab 80mg Q2W
Number analyzed (Participants) | 74 | 75
Participants | 2 | 55
Statistical Analysis 1: Comparison: Placebo vs Ixekizumab 80mg Q2W; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 102.55, 95% CI 2-sided [22.79 to 461.43]

3. Secondary Outcome: Number of Participants With at Least a 3 Point Improvement in Genital Psoriasis Itch Numeric Rating Scale (NRS) Item Within the Genital Psoriasis Symptom Scale (GPSS)
Description: GPSS is a participant-administered assessment of 8 symptoms: itch, pain, discomfort, stinging, burning, redness, scaling, and cracking. Each respondent was asked to answer the questions based on the psoriasis symptoms in his or her genital area. The overall severity for each individual genital psoriasis symptom is indicated by selecting the number from an Numeric Rating Scale (NRS) of 0 to 10 that best describes the worst level of each symptom in the genital area in the past 24 hours, where 0 (= no severity) and 10 (worst imaginable severity).
Time Frame: Week 12
Population: All randomized participants with baseline GPSS Itch NRS Score >= 3.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Ixekizumab 80mg Q2W
Number analyzed (Participants) | 60 | 62
Participants | 5 | 37
Statistical Analysis 1: Comparison: Placebo vs Ixekizumab 80mg Q2W; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 16.27, 95% CI 2-sided [5.71 to 46.40]

4. Secondary Outcome: Number of Participants Whose Frequency of Sexual Activity is Never or Rarely Limited by Genital Psoriasis, Utilizing the Genital Psoriasis Sexual Frequency Questionnaire (SFQ) Item 2
Description: The SFQ is a participant reported outcome measure to evaluate the impact of genital psoriasis symptoms on sexual frequency. It consists of 2 items that assess the impact of genital psoriasis symptoms on the frequency of sexual activity. Respondents were asked to answer the questions based on their psoriasis symptoms in the genital area. Item 2 assesses how often genital psoriasis symptoms limited the frequency of sexual activity with the following response options: 0 = never, 1 = rarely, 2 = sometimes, 3 = often, 4 = always.
  *The SFQ is also referred to as the GenPs-SFQ (genital psoriasis sexual frequency questionnaire).
Time Frame: Week 12
Population: All randomized participants with baseline GenPs-SFQ Item 2 Score >= 2.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Ixekizumab 80mg Q2W
Number analyzed (Participants) | 42 | 37
Participants | 9 | 29
Statistical Analysis 1: Comparison: Placebo vs Ixekizumab 80mg Q2W; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 13.57, 95% CI 2-sided [4.57 to 40.29]

5. Secondary Outcome: Number of Participants Whose Frequency of Avoiding Sexual Activity is Either Never or Rarely Limited by Genital Psoriasis in the Sexual Activity Avoidance Subscale Score of the Genital Psoriasis Sexual Impact Scale (GPSIS)
Description: GPSIS is a participant reported outcome measure to evaluate the impact of genital psoriasis symptoms on sexual activity.
  The GPSIS Sexual Activity Avoidance Subscale includes 2 items:
  Item 1 asks whether the participant has been sexually active in the past week. (No due to other reasons = 1, No due to genital Ps = 5) Item 2 asks how often the participant avoided sexual activity in the past week due to Genital Psoriasis. (Never = 1, rarely = 2, Sometimes = 3, Often = 4)
Time Frame: Week 12
Population: All randomized participants with baseline GPSIS sexual activity avoidance subscale score >= 3.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Ixekizumab 80mg Q2W
Number analyzed (Participants) | 35 | 30
Participants | 9 | 23
Statistical Analysis 1: Comparison: Placebo vs Ixekizumab 80mg Q2W; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 9.84, 95% CI 2-sided [3.08 to 31.40]

6. Secondary Outcome: Change From Baseline in Dermatology Life Quality Index (DLQI) Total Score
Description: DLQI is a simple, participant-administered, 10 question, validated, quality-of-life questionnaire that covers 6 domains: 1) Symptoms and feelings 2) Daily activities 3) Leisure 4) Work and school 5) Personal relationships 6) Treatment.
  Response categories include:
  0 = not at all; 1 = a little; 2 = a lot; 3 = very much; "not relevant" responses scored as "0" and total score range of 0 to 30; higher scores indicate poor quality of life.
  Least Square (LS) Mean was calculated using Mixed Model Repeated Measures (MMRM) model with treatment, baseline body surface area (BSA) category, baseline value, visit, treatment-by-visit, and baseline value-by-visit interactions as fixed effects.
Time Frame: Baseline, Week 12
Population: All randomized participants with baseline and post baseline observation for DLQI.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Ixekizumab Q2W: Participants received 160 milligrams (mg) Ixekizumab subcutaneously (SC) at baseline followed by 80 mg Ixekizumab every 2 weeks (Q2W) from week 2 to week 10. At week 12, 80 mg Ixekizumab and placebo was given SC during blinded treatment period.
Arm/Group | Placebo | Ixekizumab Q2W
Number analyzed (Participants) | 70 | 74
units on a scale | -1.4 (0.62) | -9.7 (0.59)
Statistical Analysis 1: Comparison: Placebo vs Ixekizumab Q2W; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -8.4, 95% CI 2-sided [-10.1 to -6.7], Standard Error of Mean 0.86

7. Secondary Outcome: Change From Baseline in Modified Genital Psoriasis Area and Severity Index (mGPASI) Score
Description: mGPASI determines participants psoriasis severity in the genital region at a given time point yielding an overall score of 0 for no psoriasis to 72 for the most severe disease. scoring index incorporates the degree of erythema (or redness), induration (or thickness), and scaling) of the genital plaques as well as erosion, fissure, and/or ulcer as a product of the genital area involved. LS Mean was calculated using MMRM model with treatment, baseline BSA category, baseline value, visit, treatment-by-visit, and baseline value-by-visit interactions as fixed effects.
Time Frame: Baseline, Week 12
Population: All randomized participants with baseline and post baseline observation for mGPASI.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Ixekizumab 80mg Q2W
Number analyzed (Participants) | 73 | 74
units on a scale | -3.9 (1.56) | -23.9 (1.48)
Statistical Analysis 1: Comparison: Placebo vs Ixekizumab 80mg Q2W; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -20.0, 95% CI 2-sided [-24.3 to -15.8], Standard Error of Mean 2.15

8. Secondary Outcome: Number of Participants With at Least a 2-Point Change in Patient's Global Assessment of Genital Psoriasis (PatGA-Genital)
Description: Patient's Global Assessment of Genital Psoriasis (PatGA-Genital) is a participant-administered, single-item scale on which participants are asked to rank the severity of their genital psoriasis "today" by circling a number on a 0 to 5 NRS, as follows: from 0 (clear), no genital psoriasis; to 5 (severe).
Time Frame: Week 12
Population: All randomized participants with baseline PatGA-Genital score >= 2.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Ixekizumab 80mg Q2W
Number analyzed (Participants) | 73 | 72
Participants | 11 | 51
Statistical Analysis 1: Comparison: Placebo vs Ixekizumab 80mg Q2W; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 13.95, 95% CI 2-sided [6.12 to 31.80]

9. Secondary Outcome: Change From Baseline on the Short-Form Health Survey (SF-36) Physical Component Summary (PCS)
Description: SF-36 is a participant-reported outcome measure evaluating a participant's health status. It comprises 36 items covering 8 domains: physical functioning, role physical, role emotional, bodily pain, vitality, social functioning, mental health, and general health. Items are answered on Likert scales of varying lengths. Items from 8 domains contribute to the PCS. The summary scores range from 0 to 100, with higher scores indicating better levels of function and/or better health.
  Least Squares Mean (LS Mean) was calculated using Analysis of covariance (ANCOVA) model with treatment, baseline BSA category, & baseline value and modified baseline observation carried forward (mBOCF) imputation method.
Time Frame: Baseline, Week 12
Population: All randomized participants with baseline and post baseline measurement for SF-36 PCS.
  mBOCF: Participants with or without post baseline measurement who discontinued treatment due to Adverse Event (AE) or death were imputed by their baseline observation , Participants who discontinued due to other reasons were imputed by their last observation.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Ixekizumab 80mg Q2W
Number analyzed (Participants) | 71 | 72
units on a scale | 0.687 (0.7998) | 5.193 (0.7942)
Statistical Analysis 1: Comparison: Placebo vs Ixekizumab 80mg Q2W; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Final Values) = 4.506, 95% CI 2-sided [2.264 to 6.748], Standard Error of Mean 1.1339

10. Secondary Outcome: Change From Baseline on the Short-Form Health Survey (SF-36) Mental Component Summary (MCS)
Description: SF-36 is a participant-reported outcome measure evaluating a participant's health status. It comprises 36 items covering 8 domains: physical functioning, role physical, role emotional, bodily pain, vitality, social functioning, mental health, and general health. Items are answered on Likert scales of varying lengths. Items from 8 domains contribute to the MCS. The summary scores range from 0 to 100, with higher scores indicating better levels of function and/or better health.
  Least Squares Mean (LS Mean) was calculated using Analysis of covariance (ANCOVA) model with treatment, baseline BSA category, & baseline value and modified baseline observation carried forward (mBOCF) imputation method.
Time Frame: Baseline, Week 12
Population: All randomized participants with baseline and post baseline measurement for SF-36 MCS.
  mBOCF: Participants with or without post baseline measurement who discontinued treatment due to Adverse Event (AE) or death were imputed by their baseline observation, Participants who discontinued due to other reasons were imputed by their last observation.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Ixekizumab 80mg Q2W
Number analyzed (Participants) | 71 | 72
units on a scale | 2.186 (0.7333) | 3.982 (0.7281)
Statistical Analysis 1: Comparison: Placebo vs Ixekizumab 80mg Q2W; Test type: Superiority; p = 0.085, ANCOVA; Mean Difference (Final Values) = 1.797, 95% CI 2-sided [-0.253 to 3.847], Standard Error of Mean 1.0367

11. Secondary Outcome: Change From Baseline in Genital Psoriasis Symptom Scale (GPSS) Total Score and Individual Items
Description: GPSS is a participant's-administered assessment of 8 symptoms: itch, pain, discomfort, stinging, burning, redness, scaling, and cracking. Each respondent was asked to answer the questions based on the psoriasis symptoms in his or her genital area. The overall severity for each individual genital psoriasis symptom is indicated by selecting the number from an Numeric Rating Scale (NRS) of 0 to 10 that best describes the worst level of each symptom in the genital area in the past 24 hours, where 0 (no severity) and 10 (worst imaginable severity). total score ranges from 0 (no severity) - 80 (worst imaginable severity) LS Mean was calculated using MMRM model with treatment, baseline BSA category, baseline value, visit, treatment-by-visit, and baseline value-by-visit interactions as fixed effects.
Time Frame: Baseline, Week 12
Population: All randomized participants with baseline and post baseline observation for GPSS total or individual item scores.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Ixekizumab 80mg Q2W
Number analyzed (Participants) | 66 | 69
units on a scale
  Total Score | -2.82 (2.190) | -31.57 (2.070)
  Itch | -0.21 (0.290) | -4.02 (0.274)
  Pain | -0.34 (0.294) | -3.84 (0.278)
  Discomfort | -0.42 (0.298) | -4.27 (0.282)
  Stinging | -0.51 (0.298) | -3.74 (0.281)
  Burning | -0.53 (0.289) | -3.73 (0.273)
  Redness | -0.63 (0.287) | -4.45 (0.272)
  Scaling | -0.02 (0.273) | -3.80 (0.259)
  Cracking | -0.19 (0.280) | -3.74 (0.264)
Statistical Analysis 1: Comparison: Placebo vs Ixekizumab 80mg Q2W; Total Score; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -28.75, 95% CI 2-sided [-34.72 to -22.78], Standard Error of Mean 3.015
Statistical Analysis 2: Comparison: Placebo vs Ixekizumab 80mg Q2W; Itch; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -3.81, 95% CI 2-sided [-4.60 to -3.02], Standard Error of Mean 0.399
Statistical Analysis 3: Comparison: Placebo vs Ixekizumab 80mg Q2W; Pain; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -3.50, 95% CI 2-sided [-4.30 to -2.70], Standard Error of Mean 0.405
Statistical Analysis 4: Comparison: Placebo vs Ixekizumab 80mg Q2W; Discomfort; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -3.85, 95% CI 2-sided [-4.66 to -3.04], Standard Error of Mean 0.410
Statistical Analysis 5: Comparison: Placebo vs Ixekizumab 80mg Q2W; Stinging; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -3.23, 95% CI 2-sided [-4.04 to -2.42], Standard Error of Mean 0.410
Statistical Analysis 6: Comparison: Placebo vs Ixekizumab 80mg Q2W; Burning; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -3.20, 95% CI 2-sided [-3.99 to -2.41], Standard Error of Mean 0.397
Statistical Analysis 7: Comparison: Placebo vs Ixekizumab 80mg Q2W; Redness; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -3.81, 95% CI 2-sided [-4.59 to -3.03], Standard Error of Mean 0.395
Statistical Analysis 8: Comparison: Placebo vs Ixekizumab 80mg Q2W; Scaling; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -3.78, 95% CI 2-sided [-4.53 to -3.03], Standard Error of Mean 0.377
Statistical Analysis 9: Comparison: Placebo vs Ixekizumab 80mg Q2W; Cracking; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -3.55, 95% CI 2-sided [-4.31 to -2.79], Standard Error of Mean 0.385

12. Secondary Outcome: Number of Participants Achieving sPGA of Genitalia (0,1) at Week 12 by Treatment-Emergent Anti-Drug Antibody (TE-ADA) Status and by Neutralizing Antibody (NAb) Status
Description: as for outcome 1
Time Frame: Week 12
Population: All randomized participants who received at least one dose of study drug and either had baseline and at least 1 post-baseline evaluable samples or had no evaluable baseline and all negative post-baseline anti-drug antibody negative samples.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Ixekizumab 80mg Q2W
Number analyzed (Participants) | 73 | 75
Participants
  TE-ADA positive: number analyzed (Participants) | 0 | 6
  TE-ADA positive |  | 5
  TE-ADA negative: number analyzed (Participants) | 73 | 69
  TE-ADA negative | 6 | 50
  TE-ADA inconclusive: number analyzed (Participants) | 0 | 0
  NAb positive: number analyzed (Participants) | 0 | 0
  NAb negative: number analyzed (Participants) | 0 | 0
  NAb inconclusive: number analyzed (Participants) | 0 | 6
  NAb inconclusive |  | 5

ADVERSE EVENTS:
Time Frame: Up to 667 Days
Description: Gender specific events occurring only in male or female participants have had the number of participants at risk adjusted accordingly.
Groups:
- Placebo - Blinded Treatment Period: Participants received placebo subcutaneously at baseline and every 2 weeks (Q2W) from week 2 to week 10. At week 12, 160 mg Ixekizumab was given by subcutaneous injection during blinded treatment period.
- Ixekizumab 80 mg Q2W - Blinded Treatment Period: Participants received 160 milligrams (mg) Ixekizumab subcutaneously (SC) at baseline followed by 80 mg Ixekizumab every 2 weeks (Q2W) from week 2 to week 10. At week 12, 80 mg Ixekizumab and placebo was given SC during blinded treatment period.
- Ixeqizumab 80mg Q2W - Post Treatment Follow-up Period; Ixekizumab 80mg Q4W - Post Treatment Follow-up: Participants did not receive any study treatment during post treatment follow-up period.
Arm/Group | Placebo - Blinded Treatment Period | Ixekizumab 80 mg Q2W - Blinded Treatment Period | Placebo/Ixekizumab 80mg Q4W - Open Label Treatment Period | Ixekizumab 80mg Q2W/Ixekizumab 80mg Q4W - Open Label Treatment | Placebo - Post Treatment Follow-up | Ixeqizumab 80mg Q2W - Post Treatment Follow-up Period | Ixekizumab 80mg Q4W - Post Treatment Follow-up
All-Cause Mortality (participants affected / at risk) | 0/74 | 0/75 | 0/65 | 0/74 | 0/1 | 0/49 | 0/78
Serious Adverse Events (participants affected / at risk) | 1/74 | 0/75 | 2/65 | 5/74 | 0/1 | 2/49 | 1/78
Other Adverse Events (participants affected / at risk) | 19/74 | 21/75 | 28/65 | 27/74 | 0/1 | 1/49 | 0/78
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo - Blinded Treatment Period (N=74) | Ixekizumab 80 mg Q2W - Blinded Treatment Period (N=75) | Placebo/Ixekizumab 80mg Q4W - Open Label Treatment Period (N=65) | Ixekizumab 80mg Q2W/Ixekizumab 80mg Q4W - Open Label Treatment (N=74) | Placebo - Post Treatment Follow-up (N=1) | Ixeqizumab 80mg Q2W - Post Treatment Follow-up Period (N=49) | Ixekizumab 80mg Q4W - Post Treatment Follow-up (N=78)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Escherichia bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Extradural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0/49 (0) | 1/56 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo - Blinded Treatment Period (N=74) | Ixekizumab 80 mg Q2W - Blinded Treatment Period (N=75) | Placebo/Ixekizumab 80mg Q4W - Open Label Treatment Period (N=65) | Ixekizumab 80mg Q2W/Ixekizumab 80mg Q4W - Open Label Treatment (N=74) | Placebo - Post Treatment Follow-up (N=1) | Ixeqizumab 80mg Q2W - Post Treatment Follow-up Period (N=49) | Ixekizumab 80mg Q4W - Post Treatment Follow-up (N=78)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 5 (7) | 10 (24) | 3 (6) | 0 (0) | 0 (0) | 0 (0)
Bacterial vaginosis (Infections and infestations) | 0 (0) | 0 (0) | 0/16 (0) | 1/18 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 4 (4) | 2 (2) | 9 (13) | 7 (8) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 5 (5) | 12 (12) | 10 (12) | 6 (6) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1/16 (2) | 0/18 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 0 (0) | 0 (0) | 0/16 (0) | 1/18 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 4 (6) | 3 (3) | 2 (2) | 6 (6) | 0 (0) | 0 (0) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0/16 (0) | 1/18 (1) | 0 (0) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0/16 (0) | 1/18 (1) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal discomfort (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0/0 (0) | 1/11 (1) | 0/21 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Disclosures are prohibited until after the sponsor discloses the primary and secondary publications of clinical trial data.

DOCUMENTS (4):
  • Study Protocol: Protocol (2015-11-14): https://cdn.clinicaltrials.gov/large-docs/98/NCT02718898/Prot_000.pdf
  • Study Protocol: Protocol (a) (2016-01-22): https://cdn.clinicaltrials.gov/large-docs/98/NCT02718898/Prot_001.pdf
  • Study Protocol: Protocol (b) (2016-11-22): https://cdn.clinicaltrials.gov/large-docs/98/NCT02718898/Prot_002.pdf
  • Statistical Analysis Plan (2017-03-08): https://cdn.clinicaltrials.gov/large-docs/98/NCT02718898/SAP_003.pdf